CLINICAL TRIAL: NCT02743611
Title: A Phase 1/2 Dose-Finding Study to Evaluate the Safety, Feasibility, and Activity of BPX-701, a Controllable PRAME T-Cell Receptor Therapy, in HLA-A2+ Subjects With AML, Previously Treated MDS, or Metastatic Uveal Melanoma
Brief Title: Safety & Activity of Controllable PRAME-TCR Therapy in Previously Treated AML/MDS or Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company decision
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-011
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Uveal Melanoma
Keywords: BPX-701; AP1903; rimiducid; AML; MDS; relapsed AML; uveal melanoma; PRAME
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Uveal Melanoma | interventions — AP 1903 reagent

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 Does Escalation (Experimental): Participants with relapsed AML or previously treated MDS will receive an intravenous infusion of BPX-701. Dose escalation of BPX-701 will continue until the recommended cell dose level is reached.
  Rimiducid may be administered in response to treatment-related toxicity.
  Interventions: Biological: BPX-701; Drug: Rimiducid
- Arm 2 Dose Escalation (Experimental): Participants with metastatic uveal melanoma will receive an intravenous infusion of BPX-701. Dose escalation of BPX-701 will continue until the recommended cell dose level is reached.
  Rimiducid may be administered in response to treatment-related toxicity.
  Interventions: Biological: BPX-701; Drug: Rimiducid
- Arm 1 Part 2 Dose Expansion (Experimental): Participants with relapsed AML or previously treated MDS will receive an intravenous infusion of BPX-701 at the recommended cell dose level.
  Rimiducid may be administered in response to treatment-related toxicity.
  Interventions: Biological: BPX-701; Drug: Rimiducid
- Arm 2 Part 2 Dose Expansion (Experimental): Participants with metastatic uveal melanoma will receive an intravenous infusion of BPX-701 at the recommended cell dose level.
  Rimiducid may be administered in response to treatment-related toxicity.
  Interventions: Biological: BPX-701; Drug: Rimiducid

INTERVENTIONS:
Biological: BPX-701 — autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch
Drug: Rimiducid — dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
  Other Names: AP1903

SUMMARY:
The purpose of this study is to evaluate the safety and activity of BPX-701 in participants with relapsed AML, previously treated MDS, or metastatic uveal melanoma expressing high levels of PReferentially expressed Antigen in MElanoma (PRAME). Participants' T cells are modified to recognize and target the PRAME tumor marker on cancer cells.

DETAILED DESCRIPTION:
The goal of this study is to characterize the safety, feasibility, and clinical activity of BPX-701, a genetically modified autologous T cell product incorporating an HLA-A2-restricted PRAME-directed TCR and a rimiducid-inducible safety switch, when administered to subjects with relapsed AML, previously treated MDS, or metastatic uveal melanoma.

The study will be comprised of multiple parts:

Part 1 (Phase 1): Cell dose escalation to identify the maximum dose of BPX-701 T cells (escalating doses from 1.25 x 10E6 cells/kg up to 5.0 x 10E6 cells/kg to be explored) Parts 2 and 3 (Phase 2): Dose expansion to assess the safety, pharmacodynamics (including BPX-701 T cell persistence and response to rimiducid as applicable), and clinical activity at the recommended dose identified in Part 1 During Parts 1, 2, or 3, rimiducid may be administered following BPX-701 T cell infusion in response to uncontrollable, treatment-emergent toxicity

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent
2. Participants in Arm 1:

   MDS not responding to hypomethylation therapy or recurrence after initial response AML with disease relapse following first complete remission with intermediate or adverse genetics according to the European Leukemia Net criteria. AML participants with prior stem cell transplant must be >100 days post-transplant with no evidence of active graft-versus-host disease and not requiring systemic immunomodulatory or immunosuppressive therapy (>10mg prednisone daily or treatment with a calcineurin inhibitor)
3. Participants in Arm 2:

   Metastatic uveal melanoma with a radiographically measurable tumor, absolute neutrophil count >/=1000/uL, and platelets >/=75,000/uL
4. HLA-A2.01 positive by local testing
5. Tumor with positive PRAME expression by central testing
6. Age >/= 18 years
7. Participant has a life expectancy >12 weeks and is able to carry out daily life activities without difficulty (Eastern Cooperative Oncology Group performance status 0 or 1).
8. Participant has adequate venous access for apheresis or agrees to use of a central line for blood collection.
9. Participant does not have significant side effects from previous anticancer treatment.
10. Adequate organ function including absolute lymphocyte count >/=200/uL.
11. Sexually active participants must use medically acceptable methods of contraception for at least 1 year after study treatment.

Exclusion Criteria

1. Participants with AML must not have:

   * Acute promyelocytic leukemia,
   * Primary refractory disease,
   * Uncontrolled disseminated intravascular coagulation,
   * Signs or symptoms of cancer cells in the brain or nervous system,
   * Peripheral blast count >/=20,000/uL
2. Participants with uveal melanoma must not have an untreated brain tumor
3. Participant has a history of major surgery or treatment with other cancer therapy within 2-4 weeks (1 week for hydroxyurea) before study treatment.
4. Participant has an active, autoimmune disease that requires immunosuppressive therapy. Exceptions are vitiligo, type I diabetes, certain cases of hypothyroidism and psoriasis, or Hashimoto's thyroiditis on a stable dose of thyroid replacement therapy
5. History of clinically significant heart problems.
6. Current severe, uncontrolled systemic disease including an ongoing, active infection requiring treatment with antibiotics within 2 weeks before study treatment.
7. Participant is currently pregnant or breastfeeding.
8. Participant requires chronic, systemic steroid therapy.
9. Participant is positive for Hepatitis B, Hepatitis C, HIV, syphilis, West Nile virus, or Chagas disease.
10. Participant has side effects from earlier cancer treatment that have not resolved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2020-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Contact Contact for Clinical Trials, Study Director — Bellicum Pharmaceuticals
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Oregon Health & Science University, Portland, Oregon
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Part 1: Does Escalation: Participants with relapsed AML or previously treated MDS received an intravenous infusion of BPX-701, starting at 1.25 x 10E6 cells/kg.
  This arm had planned for dose escalations of BPX-701 until the recommended cell dose levels were reached; however, each subject only received 1 dose of BPX-701. Rimiducid was planned for subjects in response to treatment-related toxicity; however, no patients in this study received rimiducid.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch
  Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
- Arm 2 Part 1: Dose Escalation: No subjects were enrolled in this arm. See below for original arm description:
  Participants with metastatic uveal melanoma will receive an intravenous infusion of BPX-701, starting at 1.5 x 10E6 cells/kg. Dose escalation of BPX-701 will continue until the recommended cell dose level is reached.
  Rimiducid may be administered in response to treatment-related toxicity.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch
  Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
- Arm 1 Part 2: Dose Expansion: No subjects were enrolled in this arm. See below for original arm description:
  Participants with relapsed AML or previously treated MDS will receive an intravenous infusion of BPX-701 at the recommended cell dose level based on Arm 1 Part 1 results.
  Rimiducid may be administered in response to treatment-related toxicity.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch
  Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
- Arm 2 Part 2: Dose Expansion: No subjects were enrolled in this arm. See below for original arm description:
  Participants with metastatic uveal melanoma will receive an intravenous infusion of BPX-701 at the recommended cell dose level based on Arm 2 Part 2 results.
  Rimiducid may be administered in response to treatment-related toxicity.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch
  Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
Period: Overall Study
Arm/Group | Arm 1 Part 1: Does Escalation | Arm 2 Part 1: Dose Escalation | Arm 1 Part 2: Dose Expansion | Arm 2 Part 2: Dose Expansion
Started (All 4 enrolled subjects were enrolled into Arm 1 and started w/ the 1.25 x 10E6 cells/kg dose.) | 4 | 0 (This study was terminated early. No subjects were enrolled in Arm 2 per Sponsor discretion.) | 0 (This study was terminated early. No subjects were enrolled in Arm 1 Part 2 per Sponsor discretion.) | 0 (This study was terminated early. No subjects were enrolled in Arm 2 Part 2 per Sponsor discretion.)
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Early study termination due to Sponsor discretion | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 Part 1: Does Escalation: Participants with relapsed AML or previously treated MDS received an intravenous infusion of BPX-701, starting at 1.25 x 10E6 cells/kg.
  This arm had planned for dose escalations of BPX-701 until the recommended cell dose levels were reached; however, each subject only received 1 dose of BPX-701. Rimiducid was planned for subjects in response to treatment-related toxicity; however, no patients in this study received rimiducid.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
  No patients were enrolled in the other 3 parts of the study due to Sponsor discretion.
Arm/Group | Arm 1 Part 1: Does Escalation
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 68.5 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Arm 1: Dose-limiting Toxicity
Description: Incidence of dose limiting-toxicity (DLT)
Time Frame: 28 days after BPX-701 infusion
Population: DLT Evaluable population: all ITT subjects in Arm 1 Part 1 who complete through Day 28 or who had a DLT during the DLT evaluation period
Measure: Count of Participants; unit: Participants
Groups:
- DLT Population: This population includes 3 of the 4 patients who participate in Arm 1 Part 1 and completed follow-up through at least 28 days following BPX-701 infusion and were thus able to be assessed for dose-limiting toxicities.
  No patients were enrolled in the other 3 parts of this study per sponsor discretion.
Arm/Group | DLT Population
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Part 1 Arm 1: Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Number of participants with AEs and SAEs assessed for severity using CTCAE
Time Frame: 15 months
Population: Subjects enrolled in Arm 1 Part 1 of the study who received the planned dose of BPX-701
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 Part 1: Dose Escalation: Participants with relapsed AML or previously treated MDS received an intravenous infusion of BPX-701, starting at 1.25 x 10E6 cells/kg.
  This arm had planned for dose escalations of BPX-701 until the recommended cell dose levels were reached; however, each subject only received 1 dose of BPX-701. Rimiducid was planned for subjects in response to treatment-related toxicity; however, no patients in this study received rimiducid.
  BPX-701: autologous T cells genetically modified to express the αβ TCR reacting with PRAME peptide/HLA-A2.01 (PRAME TCR) and an inducible safety switch Rimiducid: dimerizer infusion to activate the safety switch and induce apoptosis of the BPX-701 T cells in the event of toxicity
  No patients were enrolled in the other 3 parts of this study due to Sponsor discretion.
Arm/Group | Arm 1 Part 1: Dose Escalation
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 15 months
Description: All AEs were to be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) and assessed for severity by the Investigator using the National Cancer Institute (NCI) CTCAE v4.03. Adverse events were to be summarized by system organ class and preferred term.
Arm/Group | Arm 1 Part 1: Dose Escalation
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Part 1: Dose Escalation (N=4)
Pseudomonas bacteremia (Infections and infestations) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Neurotoxicity (Infections and infestations) | 1 (2)
Tachypnea (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Part 1: Dose Escalation (N=4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Adverse events (by preferred term) reported more than once in one or more subjects
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (8) — Adverse events (by preferred term) reported more than once in one or more subjects
Anemia (Blood and lymphatic system disorders) | 1 (6) — Adverse events (by preferred term) reported more than once in one or more subjects
Fatigue (General disorders) | 3 (3) — Adverse events (by preferred term) reported more than once in one or more subjects
Dizziness (Nervous system disorders) | 2 (3) — Adverse events (by preferred term) reported more than once in one or more subjects
Deep vein thrombosis (Vascular disorders) | 1 (3) — Adverse events (by preferred term) reported more than once in one or more subjects
Peripheral edema (General disorders) | 2 (2) — Adverse events (by preferred term) reported more than once in one or more subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02743611/Prot_SAP_000.pdf